CLINICAL TRIAL: NCT01188174
Title: Clofarabine/Ara-C Treatment Combined With Reduced-intensity Conditioning Allogeneic Stem Cell Transplantation for Acute Myeloid Leukemia in Primary Treatment Failure
Acronym: setric
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 09/6-C
Record Dates: First submitted 2010-08-11; First posted 2010-08-25 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: AML
Keywords: AML; primary induction failure
MeSH Terms: interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — The present protocol aims to test the strategy of an early Reduced Intensity Conditioning (RIC) allo-SCT; in combination with a sequential preparative regimen for allo-SCT (Clofarabine, Intermediate dose Ara-C chemotherapy, followed by RIC with Cyclophosphamide, IV Busulfan and ATG; and delayed prophylactic infusion of donor lymphocytes (DLI) will be able to improve the outcome of patients with primary treatment failure AML.

SUMMARY:
The present trial will establish a prospective sequential Allogeneic Stem Cell Transplantation (allo-SCT) treatment combining both salvage chemotherapy and Reduced Intensity Conditioning (RIC) for primary treatment failure Acute Myeloid Leukemia (AML), to which future innovative strategies can be compared.

DETAILED DESCRIPTION:
Primary Endpoint: To improve the 2 year overall survival in patients with primary treatment failure

* Secondary Endpoints:

* Feasibility of early transplantation within a multicenter trial
* Leukemia-free survival (LFS) at 2 years from transplantation
* Leukemia Response rate at day +30, +90 and 6 months
* Cumulative incidence of relapse, death from leukemia, and non-relapse mortality (NRM)
* Incidence and severity of acute and chronic Graft-versus-Host disease
* Feasibility and safety of early discontinuation of immunosuppressive therapy

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML in the status of primary induction failure (i.e. persistent leukemia after 2 courses of induction chemotherapy or persisting bone marrow hypoplasia fol-lowing induction chemotherapy +/-minimal residual disease)
* Age: 18-55 years
* Availability of an HLA identical family donor OR unrelated donor with matching in 10/10 alleles (HLA-A, B, C, DRB1, DQB1) or maximum of 1 allele or antigen mismatch OR family donor with maximum 1 allele mismatch.
* Have adequate renal and hepatic functions as indicated by the following laboratory values:
* Serum creatinine ≤1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m² as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female)
* Serum bilirubin ≤1.5 mg/dL × upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) ≤2.5 × ULN
* Alkaline phosphatase ≤2.5 × ULN

Exclusion Criteria:

* Documented chloroma
* Patients having AML M3
* Documented leukemic infiltration of CNS/cerebrospinal fluid
* Karnofsky performance score below < 60%
* Acute or chronic heart failure
* HIV infection, chronic viral hepatitis
* Severe neurological or psychiatric disorders
* Any circumstances that preclude the use of the drugs used within the protocol
* Prior allogeneic or autologous stem cell transplantation
* > 3 courses of prior chemotherapy
* Denied informed consent
* Pregnancy or denied of effective contraceptive method

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the survival rate at 2 years after transplantation | at 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, Phd, Principal Investigator — Nantes University Hospital
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHRU lille, Lille
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmette, Marseille
  - Nantes University hospital, Nantes
  - Paris saint Louis, Paris
  - CHRU de Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

REFERENCES:
- [Derived] Mohty M, Malard F, Blaise D, Milpied N, Socie G, Huynh A, Reman O, Yakoub-Agha I, Furst S, Guillaume T, Tabrizi R, Vigouroux S, Peterlin P, El-Cheikh J, Moreau P, Labopin M, Chevallier P. Sequential regimen of clofarabine, cytosine arabinoside and reduced-intensity conditioned transplantation for primary refractory acute myeloid leukemia. Haematologica. 2017 Jan;102(1):184-191. doi: 10.3324/haematol.2016.150326. Epub 2016 Aug 25. PMID 27561720